CLINICAL TRIAL: NCT02211638
Title: Blopress Tablets Special Drug Use Surveillance 「Challenge - Quality Control」
Brief Title: Candesartan Cilexetil Special Drug Use Surveillance 「Challenge - Quality Control」
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 460-017; JapicCTI-132380 (Registry Identifier: JapicCTI); JapicCTI-R171021 (Other: JapicCTI)
Record Dates: First submitted 2014-03-17; First posted 2014-08-07 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-04

CONDITIONS: Hypertension
Keywords: Drug Therapy
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Candesartan Cilexetil tablets (2 to 12 mg): Candesartan Cilexetil tablets (2 to 12 mg), orally, once daily for up to 3 months
  Interventions: Drug: Candesartan Cilexetil

INTERVENTIONS:
Drug: Candesartan Cilexetil — Candesartan Cilexetil tablet
  Other Names: Blopress

SUMMARY:
The purpose of this study is to gain an understanding of the actual use of candesartan cilexetil (Blopress) in patients with hypertension, and to examine the changes in parameters such as blood pressure.

DETAILED DESCRIPTION:
This special drug use surveillance was planned to gain an understanding of the actual use of candesartan cilexetil in the new anti-hypertensive treatment environment where angiotensin receptor blocker (ARB) combination drugs have become commercially available. The surveillance also investigated the background factors of patients continuing treatment with candesartan cilexetil and patients who switched from candesartan cilexetil to ARB combination drugs, as well as changes in parameters such as blood pressure.

The usual adult dosage of Candesartan cilexetil is 4 to 8 mg, administered orally, once daily. Meanwhile, treatment was to be started at 2 mg once daily in patients with renal impairment and the dose could be increased up to 8 mg as necessary.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients

Exclusion Criteria:

1. Inpatients
2. Patients under dialysis (planned)
3. Patients with a history of coronary artery disease/cerebrovascular disorder within 6 months
4. Patients with ≥ class III of the New York Heart Association (NYHA) classification functional classification of heart failure
5. Patients that have been prescribed with candesartan (this drug/Ecard/Unisia) in the past
6. Patients who are pregnant or may possibly become pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hypertension
Sampling Method: Non-Probability Sample
Enrollment: 18113 (Actual)
Dates: Start 2011-06-13 (Actual); Primary Completion 2013-04-25 (Actual); Study Completion 2013-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1503 investigative sites in Japan, from 13-Jun-2011 to 25-Apr-2013.
Pre-assignment Details: Participants with a diagnosis of hypertension were enrolled to receive candesartan cilexetil 4 mg - 8 mg, tablet, orally, once daily for up to the last dose of study drug (up to Month 6).
Groups:
- Candesartan Cilexetil 4 mg to 8 mg: Candesartan cilexetil 4 mg - 8 mg, tablet, orally, once daily. Meanwhile, treatment was to be started at 2 mg once daily in patients with renal impairment and the dose could be increased up to 8 mg as necessary. Participants received interventions as part of routine medical care.
Period: Overall Study
Arm/Group | Candesartan Cilexetil 4 mg to 8 mg
Started | 18113
Completed | 17130
Not Completed | 983
Not completed — Case Report Forms Uncollected | 291
Not completed — Protocol Violation | 692

BASELINE CHARACTERISTICS:
Population: Safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Candesartan Cilexetil 4 mg to 8 mg
Number analyzed (Participants) | 17130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.9 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8640
  Male | 8490
Region of Enrollment [Number; unit: Participants]
  Japan | 17130
Weight [Mean (Standard Deviation); unit: kg] | 61.3 (13.46)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 11683
  Current Smoker | 2032
  Unknown | 3415
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above. Participants may be represented in more than 1 category.
  Participants
    Had no Medical Complications | 7988
    Had Medical Complications | 9142
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above. Participants may be represented in more than 1 category.
  Participants
    Had no Medical History | 14376
    Had Medical History | 2754
Initial Dose of Study Drug [Count of Participants; unit: Participants]
  2mg/day | 528
  4mg/day | 4865
  8mg/day | 11170
  12mg/day | 556
  Other Initial Dose | 11
Concomitant Antihypertensive Drugs [Count of Participants; unit: Participants]
  Had no Concomitant Antihypertensive Drugs | 11968
  Had Concomitant Antihypertensive Drugs | 5162
Switching Antihypertensive Drugs [Count of Participants; unit: Participants]
  Had no Switching Antihypertensive Drugs | 12856
  Had Switching Antihypertensive Drugs | 4274
Status of Administration of Antihypertensive Drugs [Count of Participants; unit: Participants] — Had no Antihypertensive Drugs; Participants who had not received concomitant antihypertensive drugs and switching antihypertensive drugs prior to the start of study drug were reported. Had Antihypertensive Drugs; Participants who had received concomitant antihypertensive drugs or switching antihypertensive drugs prior to the start of study drug were reported.
  Participants
    Had no Antihypertensive Drugs | 10055
    Had Antihypertensive Drugs | 7075
Clinical Systolic Blood Pressure (SBP) (Sitting) [Mean (Standard Deviation); unit: mmHg] | 156.1 (18.67)
Clinical Diastolic Blood Pressure (DBP) (Sitting) [Mean (Standard Deviation); unit: mmHg] | 88.7 (13.47)
Early Morning Home SBP (Ave) [Mean (Standard Deviation); unit: mmHg] | 153.9 (15.89)
Early Morning Home DBP (Ave) [Mean (Standard Deviation); unit: mmHg] | 89.4 (11.41)
Evening Home SBP (Ave) [Mean (Standard Deviation); unit: mmHg] | 146.2 (15.88)
Evening Home DBP (Ave) [Mean (Standard Deviation); unit: mmHg] | 85.5 (11.59)
Spot Urine Sodium: NaS [Mean (Standard Deviation); unit: mEq/L] | 129.9 (52.78)
Spot Urine Creatinine: CrS [Mean (Standard Deviation); unit: mg/L] | 804.2 (1002.82)
Estimated 24hr Creatinine Excretion: UCr24 [Mean (Standard Deviation); unit: mg/day] — UCr24 = -2.04×age（years）＋14.89×weight（kg）＋16.14×height（cm）-2244.45
  mg/day | 1099.52 (349.732)
Estimated 24hr Sodium Excretion: UNa24 [Mean (Standard Deviation); unit: mEq/day] — UNa24 = 21.98×[(NaS/CrS) ×UCr24]^0.392
  mEq/day | 230.70 (246.267)
Salt Intake: NaCl24 [Mean (Standard Deviation); unit: g/day] — NaCl24 = UNa24×0.0585
  g/day | 13.5 (14.41)
Salt Intake: NaCl24 [Mean (Standard Deviation); unit: g/day] — NaCl24 = UNa24×0.0585 10 <= Spot Urine Sodium (mEq/L) < 500, 100 <= Spot Urine Creatinine (mg/L） < 5000
  g/day | 10.0 (2.92)
Focus on Blood Pressure (BP) Measurement [Count of Participants; unit: Participants] — Participants who were answered Home or Clinic for a question" Which blood pressure are you focusing on?" were reported.
  Participants
    Focus on Home BP than Clinic BP | 7614
    Focus on Clinic BP than Home BP | 8021
    Other | 1495

OUTCOME MEASURES:

1. Primary Outcome: Changes in Clinic Blood Pressure in the Sitting Position
Description: Changes in clinic blood pressure (systolic blood pressure -SBP and diastolic blood pressure -DBP) in the sitting position measured at Month 3, last dose of candesartan (up to Month 6) relative to baseline were reported.
Time Frame: Baseline, Month 3 and Last dose of Candesartan (up to Month 6)
Population: Safety analysis set was defined as all participants who were enrolled and completed the study. Analysis population was all participants in safety analysis set who were assessed with this outcome measure. Here 'n' is number of participants analyzed at the given timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil 4 mg to 8 mg
Number analyzed (Participants) | 16617
mmHg
  Month 3, SBP: number analyzed (Participants) | 14055
  Month 3, SBP | -20.1 (19.30)
  Last Dose of Candesartan, SBP: number analyzed (Participants) | 15211
  Last Dose of Candesartan, SBP | -18.1 (18.91)
  Month 3, DBP: number analyzed (Participants) | 14055
  Month 3, DBP | -10.4 (12.34)
  Last Dose of Candesartan, DBP: number analyzed (Participants) | 15211
  Last Dose of Candesartan, DBP | -9.3 (12.12)

2. Primary Outcome: Changes in Clinic Blood Pressure in the Sitting Position for Participants Who Continued Candesartan Therapy at Week 14
Description: Changes in clinic blood pressure (systolic blood pressure -SBP and diastolic blood pressure -DBP) in the sitting position measured at Month 3, last dose of candesartan (up to Month 6) relative to baseline in only participants who continued candesartan therapy at Week 14 were reported.
Time Frame: Baseline, Month 3 and Last dose of Candesartan (up to Month 6)
Population: Safety analysis set was defined as all participants who were enrolled and completed the study. Analysis population was participants in safety analysis set who continued candesartan therapy at Week 14 and were assessed with this outcome measure. Here 'n' is number of participants analyzed at the given timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil 4 mg to 8 mg
Number analyzed (Participants) | 11753
mmHg
  Month 3, SBP: number analyzed (Participants) | 10677
  Month 3, SBP | -19.8 (18.74)
  Last Dose of Candesartan, SBP: number analyzed (Participants) | 11677
  Last Dose of Candesartan, SBP | -19.5 (18.64)
  Month 3, DBP: number analyzed (Participants) | 10677
  Month 3, DBP | -10.1 (12.01)
  Last Dose of Candesartan, DBP: number analyzed (Participants) | 11677
  Last Dose of Candesartan, DBP | -10.0 (12.03)

3. Primary Outcome: Changes in Clinic Blood Pressure in the Sitting Position for Participants Who Switched to ARB Combination Drug Therapy at Week 14
Description: Changes in clinic blood pressure (systolic blood pressure -SBP and diastolic blood pressure -DBP) in the sitting position measured at Month 3, last dose of candesartan and last dose of ARB Combination Drug (up to Month 6) relative to baseline were reported. The data was for only participants who switched to ARB combination drug therapy from candesartan therapy at Week 14 as part of routine medical care.
Time Frame: Baseline, Month 3, Last dose of Candesartan, and Last dose of ARB Combination Drug (up to Month 6)
Population: Safety analysis set was defined as all participants who were enrolled and completed the study. Analysis population was participants in safety analysis set who switched to ARB combination drug therapy from candesartan therapy at Week 14 and were assessed with this outcome measure. Here 'n' is number of participants analyzed at the given timepoint.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil 4 mg to 8 mg
Number analyzed (Participants) | 3630
mmHg
  Month 3, SBP: number analyzed (Participants) | 3060
  Month 3, SBP | -21.7 (20.74)
  Last Dose of Candesartan, SBP: number analyzed (Participants) | 2496
  Last Dose of Candesartan, SBP | -12.3 (18.83)
  Last dose of ARB Combination Drug, SBP: number analyzed (Participants) | 3464
  Last dose of ARB Combination Drug, SBP | -26.4 (20.49)
  Month 3, DBP: number analyzed (Participants) | 3060
  Month 3, DBP | -11.8 (13.26)
  Last Dose of Candesartan, DBP: number analyzed (Participants) | 2496
  Last Dose of Candesartan, DBP | -6.4 (12.04)
  Last dose of ARB Combination Drug, DBP: number analyzed (Participants) | 3464
  Last dose of ARB Combination Drug, DBP | -14.4 (13.45)

4. Secondary Outcome: Number of Participants Who Experience at Least One Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug. Among these, events which are considered possibly associated with a medicinal product are defined as adverse drug reactions.
Time Frame: Up to Month 3
Population: Safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Candesartan Cilexetil 4 mg to 8 mg
Number analyzed (Participants) | 17130
Participants | 132

5. Primary Outcome: Changes in Clinic Blood Pressure in the Sitting Position for Participants Who Switched to Diuretic-containing ARB Combination Drug Therapy at Week 14
Description: Changes in clinic blood pressure (systolic blood pressure -SBP and diastolic blood pressure -DBP) in the sitting position measured at last dose of diuretic-containing ARB combination drug (up to Month 6) relative to baseline were reported. The data was for only participants who switched to diuretic-containing ARB combination drug therapy from candesartan therapy at Week 14 as part of routine medical care.
Time Frame: Baseline and Last dose of ARB Combination Drug (up to Month 6)
Population: Safety analysis set was defined as all participants who were enrolled and completed the study. Analysis population was participants in safety analysis set who switched to diuretic-containing ARB combination drug therapy from candesartan therapy at Week 14 and were assessed with this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil 4 mg to 8 mg
Number analyzed (Participants) | 984
mmHg
  SBP | -24.5 (20.20)
  DBP | -13.2 (13.62)

6. Primary Outcome: Changes in Clinic Blood Pressure in the Sitting Position for Participants Who Switched to Calcium Channel Blocker (CCB)-Containing ARB Combination Drug Therapy at Week 14
Description: Changes in clinic blood pressure (systolic blood pressure -SBP and diastolic blood pressure -DBP) in the sitting position measured at last dose of ARB combination drug (up to Month 6) relative to baseline were reported. The data was for only participants who switched to calcium channel blocker (CCB)-containing ARB combination drug therapy from candesartan therapy at Week 14 as part of routine medical care.
Time Frame: Baseline and Last dose of ARB Combination Drug (up to Month 6)
Population: Safety analysis set was defined as all participants who were enrolled and completed the study. Analysis population was participants in safety analysis set who switched to calcium channel blocker (CCB)-containing ARB combination drug therapy from candesartan therapy at Week 14 and were assessed with this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Candesartan Cilexetil 4 mg to 8 mg
Number analyzed (Participants) | 2666
mmHg
  SBP | -26.9 (20.54)
  DBP | -14.7 (13.53)

ADVERSE EVENTS:
Time Frame: Up to Month 3
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Participants may be represented in more than 1 category.
Arm/Group | Candesartan Cilexetil 4 mg to 8 mg
Serious Adverse Events (participants affected / at risk) | 36/17130
Other Adverse Events (participants affected / at risk) | 41/17130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan Cilexetil 4 mg to 8 mg (N=17130)
Pneumonia (Infections and infestations) | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary tumour of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Cervical myelopathy (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 2
Binocular eye movement disorder (Eye disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Mechanical ileus (Gastrointestinal disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Death (General disorders) | 1 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
Pain (General disorders) | 1
Blood bilirubin increased (Investigations) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Prostatic operation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan Cilexetil 4 mg to 8 mg (N=17130)
Dizziness (Nervous system disorders) | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.